CLINICAL TRIAL: NCT06489795
Title: A Randomized Clinical Trial Comparing Laparoscopic or Robot-assisted Radical/Simple Hysterectomy Versus Abdominal Radical/Simple Hysterectomy in Patients With Early-stage Cervical Cancer
Brief Title: German-funded Laparoscopic Approach to Cervical Cancer
Acronym: G-LACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Principal Investigator, Peter Hillemanns, Prof. Dr. med., Director Department of Gynecology and Obstetrics, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-LACC
Record Dates: First submitted 2024-06-23; First posted 2024-07-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer FIGO stage IA2; cervical cancer FIGO stage IB1; cervical cancer FIGO stage IB2; laparoscopic or robot-assisted radical/simple hysterectomy; abdominal radical/simple hysterectomy; simple hysterectomy in the case of SHAPE criteria
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Interventional, multicenter, open-label, randomized, controlled non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention: Laparoscopic or robot-assisted radical/simple hysterectomy (Experimental): In the experimental arm, patients with early-stage cervical cancer will be treated by using laparoscopic or robot-assisted radical/simple hysterectomy.
  Interventions: Procedure: Laparoscopic or robot-assisted radical/simple hysterectomy
- Control intervention: Abdominal radical/simple hysterectomy (Other): In the control arm, abdominal radical/simple hysterectomy (ARH) will be used as standard therapy.
  Interventions: Procedure: Abdominal radical/simple hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic or robot-assisted radical/simple hysterectomy — In the experimental arm, patients with early-stage cervical cancer will be treated by using laparoscopic or robot-assisted radical, or in the case of SHAPE criteria, simple hysterectomy.
  Arms: Experimental intervention: Laparoscopic or robot-assisted radical/simple hysterectomy
Procedure: Abdominal radical/simple hysterectomy — In the control arm, patients with early-stage cervical cancer will be treated by using abdominal radical, or in the case of SHAPE criteria, simple hysterectomy as standard therapy.
  Arms: Control intervention: Abdominal radical/simple hysterectomy

SUMMARY:
The G-LACC trial is a prospective, interventional, multicenter, open-label, randomized and controlled non-inferiority operative trial.

The main goal of this clinical trial is to evaluate the non-inferiority of minimally invasive radical hysterectomy in contrast to abdominal radical hysterectomy in patients with early-stage cervical cancer. In the case of SHAPE criteria, surgery may also be performed as minimally invasive or abdominal simple hysterectomy. The primary criterion for assessment is disease-free survival (DFS). As secondary outcomes, overall survival (OS), disease recurrence, quality of life, intra-/postoperative complications, and serious adverse events are recorded for assessment.

DETAILED DESCRIPTION:
Eligible patients will be randomly allocated to both treatment arms in a 1:1 ratio. Within an accrual period of 4 years, 378 patients will be included per arm (756 in total) across all sites. The Follow-up period after surgery will take a minimum of 5 years.

In the standard arm, radical hysterectomy is performed as per standard technique abdominal radical hysterectomy (Piver type 2 or 3 or Querleu & Morrow Type B or C) with salpingectomy +/- oophorectomy. Ovaries may be removed or preserved +/- transposition. Surgery includes pelvic lymph node dissection or optional sentinel lymph node biopsy (SNB) according to current guidelines in both arms.

In the experimental arm, radical hysterectomy is performed as per standard conventional 2D/3D laparoscopic or robotic assisted technique (Querleu & Morrow Type B or C) with salpingectomy +/- oophorectomy. Ovaries may be removed or preserved +/- transposition. The following protective measures are mandatory for the minimally invasive arm: LEEP/conization prior to randomization or vaginal closure prior to colpotomy. Transcervical manipulators are not permitted. Use of uterus manipulators/ cervical adapter (without transcervical device) is allowed only after LEEP/conization. Meticulous dissection of pelvic (sentinel) lymph nodes including use of endobags and avoiding the dissemination of cancer cells will be implemented (tumor hygiene).

Due to the positive results of the SHAPE trial published at Plante et al. NEJM 2024, in both arms simple hysterectomy can be considered for patients with low-risk early-stage cervical cancer (SHAPE criteria: tumor < 2 cm, < 10 mm depth of stromal invasion (LEEP/cone) BUT has to be determined BEFORE randomization. Simple hysterectomy has to be performed as extrafascial hysterectomy and the preparation of a max. 5 mm vaginal cuff is required to ensure negative margins. Surgery can be performed including removal of the sentinel lymph nodes following the concept of sentinel lymph node biopsy (SNB) and according to the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
2. Patients with FIGO stage IA2, IB1, or IB2 disease (<4 cm)
3. Patients undergoing radical hysterectomy according either to Type II or III (Piver Classification) or to Type B or C (Querleu and Morrow classification)

   OR

   Simple hysterectomy can be considered for patients with low-risk early-stage cervical cancer (SHAPE criteria: tumor < 2cm, < 10 mm depth of stromal invasion (LEEP/cone). Simple hysterectomy has to be performed as extrafascial hysterectomy and the preparation of a max. 5mm vaginal cuff is required to ensure negative margins.
4. Performance status of ECOG 0-1
5. Patient must be suitable candidates for surgery with preoperative MRI and available for assessment of serious adverse events up to one year post-surgery
6. Patients who have signed an approved Informed Consent
7. Patients with a prior malignancy only if > 5 years previous with no evidence of disease
8. Females, aged 18 years or older

Exclusion Criteria:

1. Any histology other than an adenocarcinoma, squamous cell carcinoma, or adenosquamous carcinoma of the uterine cervix
2. Tumor size of 4 cm and greater, estimated by either magnetic resonance imaging (MRI) or clinical examination
3. FIGO stage IB3 - IV
4. Patients with a history of pelvic or abdominal radiotherapy
5. Patients with evidence of metastatic disease by conventional imaging studies, enlarged pelvic or aortic lymph nodes > 2 cm, or histologically positive lymph nodes
6. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
7. Patients unable to withstand prolonged lithotomy and steep Trendelenburg position
8. Patient compliance and geographic proximity that do not allow adequate follow-up
9. Women who are pregnant
10. Patients with contraindications to surgery
11. Patients with secondary invasive neoplasm in the last 5 years (except non-melanoma skin cancer, breast cancer T1 N0 M0 grade 1 or 2 without any signs of recurrence or activity)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with operable early stage cervical cancer: International Federation of Gynecology and Obstetrics (FIGO) stage IA2 (lymph vascular invasion), IB1, or IB2 and a histologic subtype of squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma
Enrollment: 756 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | up to year 5
  Disease-free survival (DFS) is defined as the time from randomization to disease recurrence or death from any course (whichever occurs first). The date of disease recurrence is defined as the date of biopsy.

SECONDARY OUTCOMES:
Overall survival | up to year 5
  Overall survival (OS) is defined as the time from randomization to death from any cause.
Disease recurrence | up to year 5 starting 6 months post-surgery
  The date of recurrence of disease is defined as the date of biopsy. A suspicion of disease recurrence (clinical or by imaging) should be verified by histopathological assessment. Disease recurrence will be assessed and recorded at each follow-up visit starting 6 months post-surgery.
Health Related Quality of Life (HRQoL): Core questionnaire | up to year 5
  Health Related Quality of Life (HRQoL) will be assessed by using the validated questionnaire European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-30)
Health Related Quality of Life (HRQoL): Cervical cancer questionnaire | up to year 5
  Health Related Quality of Life (HRQoL) will be assessed by using the validated questionnaire EORTC QLQ Cervical Cancer Module (EORTC QLQ-CX24)
Health Related Quality of Life (HRQoL): General health status | up to year 5
  Health Related Quality of Life (HRQoL) will be assessed by using the validated questionnaire EuroQoL EQ-5D-3L
Health Related Quality of Life (HRQoL): Sexual activity | up to year 5
  Health Related Quality of Life (HRQoL) will be assessed by using the validated sexual activity questionnaires (SAQ).
Lymphatic side effects: Investigator assessment | up to year 5
  Lymphatic side effects will be assessed by the investigator using Common Terminology Criteria for Adverse Events (CTCAE 3.0)
Lymphatic side effects: Patient assessment | up to year 5
  Lymphatic side effects will be assessed by the patient using the Lymphoedema Quality-of-Life (LYMQOL) questionnaire.
Complications and treatment-associated morbidity | up to one year after surgery
  Treatment-related intraoperative complications are recorded on the day of surgery according to Rosenthal's definition.
  Treatment-related postoperative complications are recorded from the day of surgery until one year after surgery.
Serious adverse events | up to one year after surgery
  Serious adverse events (SAEs) will be captured from the day of surgery until one year post surgery. Treatment-related SAEs are documented as intra-/postoperative complications according to Outcome 5.
Health care costs: Cost-effectiveness | up to year 5
  Cost-effectiveness will be determined as incremental cost-effectiveness ratios.
Health care costs: Direct cost assessment | up to year 5
  Direct costs will be assessed via internal accounting and billing systems within the hospitals.
Health care costs: Cost-utility analysis | up to year 5
  Quality-adjusted life years (QALY) calculations will be used for a cost-utility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillemanns, Prof. Dr., Principal Investigator — Hannover Medical School, Department of Gynecology and Obstetrics
Locations (14):
- Germany (14):
  - Ludwigsburg Hospital, Department of Gynecology and Obstetrics, Ludwigsburg, Baden-Wurttemberg
  - University Medical Center Tübingen, Department of Gynecology, Tübingen, Baden-Wurttemberg
  - Hochtaunus-Clinics Bad Homburg, Department of Gynecology, Bad Homburg, Hesse
  - University Medical Center Göttingen, Department of Gynecology and Obstetrics, Göttingen, Lower Saxony
  - Hannover Medical School, Department of Gynecology and Obstetrics, Hanover, Lower Saxony
  - Hospital Lüneburg, Department of Gynecology, Lüneburg, Lower Saxony
  - Hospital Bielefeld - Center, Department of Gynecology, Bielefeld, North Rhine-Westphalia
  - University Medical Center Düsseldorf, Department of Gynecology and Obstetrics, Düsseldorf, North Rhine-Westphalia
  - Protestant Hospital Wesel, Gynecological Cancer Center, Wesel, North Rhine-Westphalia
  - University Medical Center Mainz, Department of Obstetrics and Gynecology, Mainz, Rhineland-Palatinate
  - University Hospital Schleswig-Holstein, Campus Kiel, Department of Gynecology and Obstetrics, Kiel, Schleswig-Holstein
  - Vivantes Auguste-Viktoria-Hospital, Department of Gynecology, Berlin Schöneberg, State of Berlin
  - Martin Luther Hospital Berlin, Department of Gynecology and Obstetrics, Berlin
  - University Medical Center Hamburg-Eppendorf, Department of Gynecology, Hamburg